CLINICAL TRIAL: NCT06960434
Title: Systemic Interpretation of Personal and Environmental Characteristics in Overweight and Obesity: From Data Patterns to Practical Interventions
Brief Title: Mapping Obesity-related Subtypes And Interconnected Clusters
Acronym: MOSAIC
Status: Not yet recruiting | Type: Observational
Sponsor: Zuyd University of Applied Sciences (Other)
Collaborators: Statistics Netherlands (CBS) (Unknown); LIME Limburg Measures (Unknown)
Responsible Party: Sponsor
Other Study IDs: Overweight_SHICLIME_2025
Record Dates: First submitted 2025-04-14; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Overweight (BMI > 25)
Keywords: overweight; obesity; prevention; lifestyle; data-driven; clusters
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the Netherlands, about half of all adults are currently living with overweight. This number is expected to rise to as much as 64% by the year 2050, especially among younger adults aged 18 to 44. Overweight and obesity increase the risk of chronic conditions such as heart disease, diabetes, and joint problems. However, there is no single cause behind these issues. Instead, they result from a complex combination of factors - including nutrition, physical activity, sleep, stress, income, environment, and even air quality. These factors often influence each other and vary from person to person.

This study aims to better understand these patterns and connections. By analyzing large sets of data, researchers are identifying different subtypes of people with overweight or obesity. These subtypes reflect groups of individuals who share similar personal, lifestyle, and environmental characteristics. Understanding these differences makes it possible to develop more personalized lifestyle advice and support. That way, care and prevention efforts can be better tailored to what people actually need and what works best for them in practice. Experts from various fields are helping interpret the results, so that scientific insights can be translated into practical solutions for individuals, communities, and healthcare settings.

DETAILED DESCRIPTION:
Overweight and obesity are increasingly prevalent in the Netherlands. Obesity-related health issues are complex and influenced by multiple interacting variables, including personal behaviors, socioeconomic status, environmental characteristics, and health conditions. This study seeks to validate and enrich the results of an ongoing exploratory data analysis by involving experts in the interpretation of identified factor clusters related to BMI categories.

This mixed methods study includes a quantitative component (an online survey) and a qualitative component (expert panel group discussions). Experts are recruited through purposive and snowball sampling and participate in interpreting variable clusters, assessing associations, and drawing conclusions on implications for further research and practical application.

ELIGIBILITY:
Inclusion Criteria:

* researchers or professionals with expertise in obesity, lifestyle, environment, psychosocial or medical factors;
* experience in data interpretation and/or public health;
* able to communicate in Dutch;
* willing to participate in the online survey and/or expert panel meeting

Exclusion Criteria:

* no relevant domain expertise;
* inability to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of expert researchers and professionals from diverse domains including obesity research, medical and psychosocial health, lifestyle behavior, and environmental health sciences. Participants are selected using purposive sampling within the professional networks of the research team, followed by snowball sampling to include additional relevant experts. All participants have demonstrable expertise in interpreting data related to BMI or related influencing factors, and are capable of contributing to the interpretation of complex variable clusters from an interdisciplinary perspective.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Expert-perceived relationships between identified factors and BMI and expert assessment on identified data-clusters. | Baseline
  A self-developed questionnaire will be used to investigate and describe expert opinions on (1) the perceived relationsships between specific factors and BMI and (2) the expert assessment regarding data-clusters within BMI categories that has been identified in a previous study. First, the experts are invited to respond to the following question "Do you recognise a relationship between these characteristics and BMI?" on a 3-point likert scale: (1) No, I see absolutely nog relationship. (2) Yes, there may be a relationship, (3) Ik do not know. There will be space for a note. Second, identified data-clusters will be described. The experts are invited to give a brief interpretation of these clusters from their own area of expertise in an open question.

SECONDARY OUTCOMES:
Expert interpretation of within-cluster relationships and inter-cluster differences | One week after baseline
  An expert panel focus group discussion will be organized using different co-creation methods to further explore on the data-clusters within the BMI categories. By having experts from different fields share knowledge and interpretations, we expect to arrive at descriptions of specific subgroups within different BMI categories and about implications for further research and clinical implications (qualitative data-analysis).

IPD SHARING:
Plan to Share IPD: Undecided